CLINICAL TRIAL: NCT04568603
Title: A Clinical Trial to Study the Effect of a Single Dose of Islatravir (MK-8591) on the Pharmacokinetics of Methadone
Brief Title: Islatravir and Methadone Pharmacokinetics (MK-8591-029)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 8591-029; MK-8591-029 (Other: MSD Protocol Number)
Record Dates: First submitted 2020-09-23; First posted 2020-09-29 (Actual); Results first posted 2023-12-11 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — islatravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Methadone + ISL (Experimental): Methadone-maintained participants (20 to 200 mg [locally-provided] once daily [QD] from Day -14 to Day -1 and Day 10 to Day 15) receive methadone 20 to 200 mg QD on Day 1 to Day 9; ISL 60 mg is co-administered with methadone on Day 2.
  Interventions: Drug: Islatravir

INTERVENTIONS:
Drug: Islatravir — ISL 30 mg x 2 (60 mg total) capsules taken by mouth.
  Other Names: MK-8591

SUMMARY:
The present study is designed to determine the effect of islatravir (ISL) [MK-8591] on methadone pharmacokinetics (PK). The primary objective is to assess whether ISL impacts the area under the plasma concentration time curve from dosing to 24 hours postdose (AUC0-24) of S-methadone and R-methadone in participants on oral methadone therapy. It is hypothesized that the plasma AUC0-24hr for S- and R-methadone will be similar after methadone alone compared to methadone and ISL 60 mg coadministration.

ELIGIBILITY:
Inclusion Criteria:

* Has a body mass index (BMI) > 18 and ≤ 35 kg/m^2
* Is in good health based on laboratory safety tests obtained at the screening visit and prior to administration of study drug
* Is in good health based on medical history, physical examination, vital sign measurements, and electrocardiograms (ECGs) performed prior to randomization.
* Has a negative human immunodeficiency virus (HIV) antigen/antibody test at screening
* For male participants, follows contraception guidance consistent with local regulations
* For female participants:
* Is not a woman of childbearing potential (WOCBP) or
* Is a WOCBP and using acceptable contraception or is abstinent
* Is reliably participating in a methadone maintenance program for at least two (2) months prior to Day 1
* Agrees to not change their current maintenance methadone dose of 20-200 mg administered as a single daily dose

Exclusion Criteria:

* Has a history of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases
* Is mentally or legally incapacitated, has significant emotional problems at the time of prestudy (screening) visit or expected during the conduct of the study or has a history of clinically significant psychiatric disorder of the last 5 years
* Has a history of cancer (malignancy)
* Has a history of significant multiple and/or severe allergies (eg, food, drug, latex) or has had an anaphylactic reaction or significant intolerability (ie, systemic allergic reaction) to prescription or non-prescription drugs or food
* Had major surgery, donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks prior to the screening visit
* With the exception of methadone, is unable to refrain from or anticipates the use of any medication, including prescription and non-prescription drugs or herbal remedies beginning approximately 2 weeks (or 5 half-lives) prior to the first dose of the 14-day methadone maintenance run-in phase prior to Day 1, throughout the trial, until the AE follow-up call (Day 16)
* Has participated in another investigational study within 4 weeks (or 5 half-lives) prior to the prestudy (screening) visit.
* Has a QTc interval >450 msec (males) or >470 msec (females), has a history of risk factors for Torsades de Pointes (eg, heart failure/cardiomyopathy or family history of long QT syndrome), has uncorrected hypokalemia or hypomagnesemia, is taking concomitant medications that prolong the QT/QTc interval other than methadone
* Does not limit smoking to no more than 10 cigarettes per day while in the clinical research unit (CRU)
* Consumes greater than 3 glasses of alcoholic beverages per day
* Consumes excessive amounts, defined as greater than 6 servings (1 serving is approximately equivalent to 120 mg of caffeine) of coffee, tea, cola, energy drinks, or other caffeinated beverages per day
* With the exception of tetrahydrocannabinol (THC), has a positive screen for drugs with a high potential for abuse such as cocaine, amphetamines, methylenedioxymethamphetamine (MDMA), barbiturates, benzodiazepines (with the exception noted in exclusion criteria 7), or opiates/opioids on Day -1
* Presents any concern by the investigator regarding safe participation in the study or for any other reason the investigator considers the participant inappropriate for participation in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2021-07-09 (Actual); Study Completion 2021-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (2):
- United States (2):
  - Research Centers of America, LLC ( Site 0002), Hollywood, Florida
  - PRA Health Sciences ( Site 0001), Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Matthews RP, Ankrom W, Handy W, Patel M, Matthews C, Xu Z, Gravesande K, Searle S, Schwartz H, Stoch SA, Iwamoto M. A Phase 1 Study to Evaluate the Pharmacokinetic Drug-Drug Interaction Between Islatravir and Methadone in Participants on Stable Methadone Therapy. Clin Pharmacol Drug Dev. 2025 Jan;14(1):36-43. doi: 10.1002/cpdd.1492. Epub 2024 Dec 8. PMID 39648614

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Methadone-maintained participants were recruited at 2 study sites in the United States.
Groups:
- Methadone + ISL: Methadone-maintained participants (20 to 200 mg [locally-provided] once daily [QD] from Day -14 to Day -1) receive their usual methadone dose on Day 1 and Days 3 to 14. On Day 2, methadone is coadministered with islatravir (ISL) 60 mg.
Period: Overall Study
Arm/Group | Methadone + ISL
Started | 14
Received ISL on Day 2 | 13
Completed | 13
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Groups:
- Methadone + ISL: Methadone-maintained participants (20 to 200 mg [locally-provided] QD from Day -14 to Day -1) receive their usual methadone dose on Day 1 and Days 3 to 14. On Day 2, methadone is coadministered with ISL 60 mg.
Arm/Group | Methadone + ISL
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.5 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 12
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Dose-Normalized Area Under the Plasma Concentration Time Curve From 0-24 Hours Postdose (AUC0-24) of R-Methadone
Description: The AUC0-24 of R-methadone was determined on Day 1 (methadone) and Day 2 (methadone + ISL). Back-transformed least-squares mean and confidence interval from mixed effects model were performed on natural log-transformed values; data show the geometric least squares mean.
Time Frame: Days 1 and 2: predose and 0.5, 1, 1.5, 2, 3, 4, 6, 12, 16, and 24 hours postdose
Population: All participants who complied with the protocol sufficiently to ensure that generated data were likely to exhibit the effects of treatment, according to the underlying scientific model, are included.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ng*h/mL/mg
Arm/Group | Methadone + ISL
Number analyzed (Participants) | 13
ng*h/mL/mg
  Day 1: Methadone Alone | 61.9 [49.3 to 77.7]
  Day 2: Methadone + ISL | 63.9 [52.2 to 78.1]
Statistical Analysis 1: Comparison: Methadone + ISL; Test type: Equivalence — The hypothesis that administration of methadone + ISL is similar to the methadone alone will be supported if the 90% CI for the geometric mean ratio (GMR) of methadone+ ISL to methadone alone is contained within the interval (0.70, 1.43); GMR = 1.03, 90% CI 2-sided [1.00 to 1.07]

2. Primary Outcome: Dose-Normalized AUC0-24 of S-Methadone
Description: The AUC0-24hr of S-methadone was determined on Day 1 (methadone) and Day 2 (methadone + ISL). Back-transformed least-squares mean and confidence interval from mixed effects model were performed on natural log-transformed values; data show the geometric least squares mean.
Time Frame: Days 1 and 2: predose and 0.5, 1, 1.5, 2, 3, 4, 6, 12, 16, and 24 hours postdose
Population: as for outcome 1
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ng*h/mL/mg
Groups:
- Methadone + ISL: Methadone-maintained participants (20 to 200 mg [locally-provided] once daily [QD] from Day -14 to Day -1) receive their usual methadone dose on Day 1 and Days 3 to 14. On Day 2, methadone is coadministered with ISL 60 mg.
Arm/Group | Methadone + ISL
Number analyzed (Participants) | 13
ng*h/mL/mg
  Day 1: Methadone Alone | 63.1 [48.9 to 81.5]
  Day 2: Methadone + ISL | 65.1 [51.7 to 82.0]
Statistical Analysis 1: Comparison: Methadone + ISL; Test type: Equivalence — The hypothesis that administration of methadone + ISL is similar to the methadone alone will be supported if the upper bound of the 90% CI for the GMR of methadone+ ISL to methadone alone is below 2.0; GMR = 1.03, 90% CI 2-sided [0.99 to 1.07]

3. Secondary Outcome: Dose-Normalized Maximum Plasma Concentration (Cmax) of R-Methadone
Description: The Cmax of R-methadone was determined on Day 1 (methadone) and Day 2 (methadone + ISL). Back-transformed least-squares mean and confidence interval from mixed effects model were performed on natural log-transformed values; data show the geometric least squares mean.
Time Frame: Days 1 and 2: predose and 0.5, 1, 1.5, 2, 3, 4, 6, 12, 16, and 24 hours postdose
Population: as for outcome 1
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ng/mL/mg
Arm/Group | Methadone + ISL
Number analyzed (Participants) | 13
ng/mL/mg
  Day 1: Methadone Alone | 3.64 [3.00 to 4.43]
  Day 2: Methadone + ISL | 3.71 [3.14 to 4.40]
Statistical Analysis 1: Comparison: Methadone + ISL; Test type: Equivalence — The hypothesis that administration of methadone + ISL is similar to the methadone alone will be supported if the upper bound of the 90% CI for the GMR of methadone+ ISL to methadone alone is below 1.43; GMR = 1.02, 90% CI 2-sided [0.96 to 1.09]

4. Secondary Outcome: Dose-Normalized Plasma Concentration 24 Hours Postdose (C24) of R-Methadone
Description: The C24 of R-methadone was determined on Day 1 (methadone) and Day 2 (methadone + ISL). Back-transformed least-squares mean and confidence interval from mixed effects model were performed on natural log-transformed values; data show the geometric least squares mean.
Time Frame: Days 1 and 2: 24 hours postdose
Population: as for outcome 1
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ng/ml/mg
Arm/Group | Methadone + ISL
Number analyzed (Participants) | 13
ng/ml/mg
  Day 1: Methadone Alone | 2.09 [1.63 to 2.69]
  Day 2: Methadone + ISL | 2.23 [1.78 to 2.78]
Statistical Analysis 1: Comparison: Methadone + ISL; Test type: Equivalence — The hypothesis that administration of methadone + ISL is similar to methadone alone will be supported if the upper bound of the 90% CI for the GMR of methadone+ ISL to methadone alone is below 2.0; GMR = 1.06, 90% CI 2-sided [1.03 to 1.10]

5. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of R-Methadone
Description: The Tmax of R-methadone was determined on Day 1 (methadone) and Day 2 (methadone + ISL).
Time Frame: Days 1 and 2: predose and 0.5, 1, 1.5, 2, 3, 4, 6, 12, 16, and 24 hours postdose
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Methadone + ISL
Number analyzed (Participants) | 13
hours
  Day 1: Methadone Alone | 2.00 [1.47 to 3.00]
  Day 2: Methadone + ISL | 2.00 [0.67 to 4.00]

6. Secondary Outcome: Dose-Normalized Cmax of S-Methadone
Description: The Cmax of S-methadone was determined on Day 1 (methadone) and Day 2 (methadone + ISL). Back-transformed least-squares mean and confidence interval from mixed effects model were performed on natural log-transformed values; data show the geometric least squares mean.
Time Frame: Days 1 and 2: predose and 0.5, 1, 1.5, 2, 3, 4, 6, 12, 16, and 24 hours postdose
Population: as for outcome 1
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ng/mL/mg
Arm/Group | Methadone + ISL
Number analyzed (Participants) | 13
ng/mL/mg
  Day 1: Methadone Alone | 4.25 [3.45 to 5.25]
  Day 2: Methadone + ISL | 4.31 [3.49 to 5.32]
Statistical Analysis 1: Comparison: Methadone + ISL; Test type: Equivalence — [test comment as in outcome 4, analysis 1]; GMR = 1.01, 90% CI 2-sided [0.94 to 1.09]

7. Secondary Outcome: Dose-Normalized C24 of S-Methadone
Description: The C24 of S-methadone was determined on Day 1 (methadone) and Day 2 (methadone + ISL). Back-transformed least-squares mean and confidence interval from mixed effects model were performed on natural log-transformed values; data show the geometric least squares mean.
Time Frame: Days 1 and 2: 24 hours postdose
Population: as for outcome 1
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ng/ml/mg
Arm/Group | Methadone + ISL
Number analyzed (Participants) | 13
ng/ml/mg
  Day 1: Methadone Alone | 1.91 [1.44 to 2.54]
  Day 2: Methadone + ISL | 2.07 [1.60 to 2.68]
Statistical Analysis 1: Comparison: Methadone + ISL; Test type: Equivalence — [test comment as in outcome 4, analysis 1]; GMR = 1.08, 90% CI 2-sided [1.04 to 1.13]

8. Secondary Outcome: Tmax of S-Methadone
Description: The Tmax of S-methadone was determined on Day 1 (methadone) and Day 2 (methadone + ISL).
Time Frame: Days 1 and 2: predose and 0.5, 1, 1.5, 2, 3, 4, 6, 12, 16, and 24 hours postdose
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Methadone + ISL
Number analyzed (Participants) | 13
hours
  Day 1: Methadone Alone | 1.50 [1.02 to 3.00]
  Day 2:Methadone + ISL | 2.00 [0.67 to 3.00]

9. Secondary Outcome: Dose-Normalized AUC0-24 of Total Methadone
Description: The AUC0-24hr of total methadone was determined on Day 1 (methadone) and Day 2 (methadone + ISL). Back-transformed least-squares mean and confidence interval from mixed effects model were performed on natural log-transformed values; data show the geometric least squares mean.
Time Frame: Days 1 and 2: predose and 0.5, 1, 1.5, 2, 3, 4, 6, 12, 16, and 24 hours postdose
Population: as for outcome 1
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ng*h/mL/mg
Arm/Group | Methadone + ISL
Number analyzed (Participants) | 13
ng*h/mL/mg
  Day 1: Methadone Alone | 126 [99.1 to 159]
  Day 2: Methadone + ISL | 129 [105 to 160]
Statistical Analysis 1: Comparison: Methadone + ISL; Test type: Equivalence — [test comment as in outcome 4, analysis 1]; GMR = 1.03, 90% CI 2-sided [0.99 to 1.07]

10. Secondary Outcome: Dose-Normalized Cmax of Total Methadone
Description: The Cmax of total methadone was determined on Day 1 (methadone) and Day 2 (methadone + ISL). Back-transformed least-squares mean and confidence interval from mixed effects model were performed on natural log-transformed values; data show the geometric least squares mean.
Time Frame: Days 1 and 2: predose and 0.5, 1, 1.5, 2, 3, 4, 6, 12, 16, and 24 hours postdose
Population: as for outcome 1
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ng/mL/mg
Arm/Group | Methadone + ISL
Number analyzed (Participants) | 13
ng/mL/mg
  Day 1: Methadone Alone | 7.91 [6.48 to 9.66]
  Day 2: Methadone + ISL | 8.02 [6.64 to 9.68]
Statistical Analysis 1: Comparison: Methadone + ISL; Test type: Equivalence — [test comment as in outcome 4, analysis 1]; GMR = 1.01, 90% CI 2-sided [0.95 to 1.08]

11. Secondary Outcome: Dose-Normalized C24 of Total Methadone
Description: The C24 of total methadone was determined on Day 1 (methadone) and Day 2 (methadone + ISL). Back-transformed least-squares mean and confidence interval from mixed effects model were performed on natural log-transformed values; data show the geometric least squares mean.
Time Frame: Days 1 and 2: 24 hours postdose
Population: as for outcome 1
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ng/ml/mg
Arm/Group | Methadone + ISL
Number analyzed (Participants) | 13
ng/ml/mg
  Day 1: Methadone Alone | 4.03 [3.10 to 5.23]
  Day 2: Methadone + ISL | 4.32 [3.42 to 5.45]
Statistical Analysis 1: Comparison: Methadone + ISL; Test type: Equivalence — [test comment as in outcome 4, analysis 1]; GMR = 1.07, 90% CI 2-sided [1.03 to 1.11]

12. Secondary Outcome: Tmax of Total Methadone
Description: The Tmax of total methadone was determined on Day 1 (methadone) and Day 2 (methadone + ISL).
Time Frame: Days 1 and 2: predose and 0.5, 1, 1.5, 2, 3, 4, 6, 12, 16, and 24 hours postdose
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Methadone + ISL
Number analyzed (Participants) | 13
hours
  Day 1: Methadone Alone | 2.00 [1.47 to 3.00]
  Day 2: Methadone + ISL | 2.00 [0.67 to 3.00]

13. Secondary Outcome: Number of Participants With Adverse Events (AEs) Following Methadone + ISL Coadministration
Description: The number of participants with AEs will be determined for 14 days after coadministration of methadone and ISL on Day 2.
Time Frame: Up to 16 days
Population: All participants who received ISL on Day 2 are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Methadone + ISL
Number analyzed (Participants) | 13
Participants | 4

14. Secondary Outcome: Number of Participants Discontinuing Study Therapy Due to AEs Following Coadministration of Methadone and ISL
Description: The number of participants discontinuing study therapy due to AEs after methadone + ISL on Day 2 will be determined.
Time Frame: Up to 15 days
Population: All participants who received ISL on Day 2 are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Methadone + ISL
Number analyzed (Participants) | 13
Participants | 0

ADVERSE EVENTS:
Time Frame: Up to 16 days (up to 14 days after methadone + ISL coadministration on Day 2)
Description: All enrolled study participants are included in analysis of all-cause mortality. All participants who received ISL on Day 2 are included in analysis of serious AEs (SAEs) and nonserious AEs.
Arm/Group | Methadone + ISL
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 4/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Methadone + ISL (N=14)
Vomiting (Gastrointestinal disorders) | 1
Infusion site extravasation (General disorders) | 1
Increased appetite (Metabolism and nutrition disorders) | 2
Headache (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 1
Nightmare (Psychiatric disorders) | 1
Papule (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-28): https://cdn.clinicaltrials.gov/large-docs/03/NCT04568603/Prot_SAP_000.pdf